CLINICAL TRIAL: NCT06205316
Title: Randomized Phase III Trial of SBRT Versus Hypofractionated Radiotherapy for Salvage of Biochemically Recurrent or Oligometastatic Prostate Adenocarcinoma After Radical Prostatectomy
Brief Title: SBRT Versus Hypofractionated Radiotherapy for Biochemically Recurrent or Oligometastatic Prostate Adenocarcinoma
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GMROA2255; NCI-2023-10897 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-009244 (Other: Mayo Clinic Institutional Review Board); GMROA2255 (Other: Mayo Clinic in Arizona)
Record Dates: First submitted 2024-01-04; First posted 2024-01-16 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Biochemically Recurrent Prostate Carcinoma; Oligometastatic Prostate Carcinoma; Recurrent Prostate Adenocarcinoma; Stage IIB Prostate Cancer AJCC v8; Stage IIC Prostate Cancer AJCC v8; Stage III Prostate Cancer AJCC v8; Stage IV Prostate Cancer AJCC v8
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Androgen Antagonists; Specimen Handling; Radiation Dose Hypofractionation; Radiation; Magnetic Resonance Spectroscopy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group I (SBRT) (Experimental): Patients undergo SBRT over 15-20 minutes every other day for a total of 5 treatments over 1-2 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive androgen deprivation therapy for up to 18 months, as clinically indicated. Patients undergo PET at screening and treatment failure, and blood sample collection throughout the study. Patients may also undergo MRI as clinically indicated at screening and treatment failure.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Biospecimen Collection; Procedure: Positron Emission Tomography; Radiation: Stereotactic Body Radiation Therapy; Other: Survey Administration; Procedure: Magnetic Resonance Imaging
- Group II (Hypofractionated radiation therapy) (Experimental): Patients undergo hypofractionated radiation therapy over 15-20 minutes once per day for a total of 20 treatments over 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive androgen deprivation therapy for up to 18 months, as clinically indicated. Patients undergo PET at screening and treatment failure, and undergo blood sample collection throughout the study. Patients may also undergo MRI as clinically indicated at screening and treatment failure.
  Interventions: Drug: Antiandrogen Therapy; Procedure: Biospecimen Collection; Radiation: Hypofractionated Radiation Therapy; Procedure: Positron Emission Tomography; Other: Survey Administration; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Drug: Antiandrogen Therapy — Receive ADT
  Other Names: ADT; Androgen Deprivation Therapy; Androgen Deprivation Therapy (ADT); Anti-androgen Therapy; Anti-androgen Treatment; Antiandrogen Treatment; Hormone Deprivation Therapy; Hormone-Deprivation Therapy
Procedure: Biospecimen Collection — Undergo blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Radiation: Hypofractionated Radiation Therapy — Undergo hypofractionated radiation therapy
  Other Names: Hypofractionated; Hypofractionated Radiotherapy; hypofractionation; Radiation, Hypofractionated
  Arms: Group II (Hypofractionated radiation therapy)
Procedure: Positron Emission Tomography — Undergo PET scan
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; proton magnetic resonance spectroscopic imaging; PT
Radiation: Stereotactic Body Radiation Therapy — Undergo SBRT
  Other Names: SABR; SBRT; Stereotactic Ablative Body Radiation Therapy
  Arms: Group I (SBRT)
Other: Survey Administration — Ancillary study
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance Imaging (MRI); MRI; Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; Structural MRI; sMRI; nuclear magnetic resonance imaging; NMRI; NMR Imaging; MRI Scan; MRIs

SUMMARY:
This phase III trial tests the side effects of stereotactic body radiation therapy (SBRT) compared to hypofractionated radiotherapy for treating patients with prostate adenocarcinoma that has come back after a period of improvement (recurrent) or that has spread from where it first started (primary site) to a limited number of sites (oligometastatic). SBRT is a type of external radiation therapy that uses special equipment to position a patient and precisely deliver radiation to tumors in the body (except the brain). The total dose of radiation is divided into smaller doses given over several days. This type of radiation therapy helps spare normal tissue. Hypofractionated radiation therapy delivers higher doses of radiation therapy over a shorter period of time and may kill more tumors cells and have fewer side effects. SBRT may work just as well as hypofractionated radiation therapy at treating patients with biochemically recurrent or oligometastatic prostate cancer, but with a shorter treatment time and possibly fewer side effects.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if salvage SBRT is non-inferior to moderately hypofractionated radiation therapy regarding treatment related rates of genitourinary (GU) and gastrointestinal (GI) grade 3 or higher within 2-years.

EXPLORATORY OBJECTIVES:

I. After completion of radiation therapy, determine the incidence of:

Ia. Disease free survival (DFS), defined as the first occurrence of new clinical failure (local recurrence, regional recurrence, or distant metastasis) after salvage radiation therapy (RT); Ib. Grade 2 or greater GU and GI toxicity at 3 years [Common Terminology Criteria for Adverse Events (CTCAE) version 5]; Ic. Grade 3 or greater GU and GI toxicity at 3 years (CTCAE version 5); Id. Quality of life following completion of radiation therapy; Ie. Impotence after the use of radiation therapy at 3 years; If. Freedom from biochemical failure (FFBF) at 5 years; Ig. Local failure at 5 years; Ih. Regional failure at 5 years; Ii. Distant failure at 5 years; Ij. Salvage androgen deprivation therapy (ADT) use (SAD) at 5 years; Ik. Progression free survival: using clinical, biochemical and SAD as events at 5 years; Il. Overall survival at 5 years; Im. Disease-specific survival at 5 years. II. Determine the impact of salvage SBRT and hypofractionated radiation therapy (HFRT) on quality of life.

III. Determine prostate and normal structure movement during RT with the use of scans.

IV. Correlate pathologic and radiologic findings with outcomes. V. Correlate pre-RT prostate specific antigen (PSA) levels with outcomes. VI. Prospectively collect information that will help to define dose-volume relationships of normal structures with acute and chronic toxicity.

VII. Allow for future research of pathologic risk factors that may influence prognosis; this information will help us to attempt to characterize their presence in prostate cancer with high-risk features after prostatectomy and their potential effect on outcomes.

VIII. Prospectively record contours that were manually drawn versus (vs.) edited from artificial intelligence (AI)-generated contours.

IX. Determine the impact of using artificial intelligence (AI) tools for automatic segmenting prostate bed and other organs at risk, in terms of toxicities and outcome.

X. Determine if there are any significant differences in dose-volumes results for cases that involved AI-autosegmentation vs. cases without.

XI. Determine the relationship between the use of AI-autosegmentation tools with toxicities and outcome.

XII. Different online daily imaging guidance systems are allowed in this trial, including x-rays, conventional Feldkamp-Davis-Kress (FDK)-based cone beam computed tomography (CBCT), and iterative CBCT. Subgroup analysis will be performed to determine patient alignment accuracy and toxicities rates with respect to different online daily imaging systems.

OUTLINE: Patients are randomized to 1 of 2 groups.

GROUP I: Patients undergo SBRT over 15-20 minutes every other day for a total of 5 treatments over 1-2 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive androgen deprivation therapy for up to 18 months, as clinically indicated. Patients undergo positron emission tomography (PET) at screening and treatment failure, and blood sample collection throughout the study. Patients may also undergo magnetic resonance imaging (MRI) as clinically indicated at screening and treatment failure.

GROUP II: Patients undergo hypofractionated radiation therapy over 15-20 minutes once per day for a total of 20 treatments over 4-6 weeks in the absence of disease progression or unacceptable toxicity. Patients may receive androgen deprivation therapy for up to 18 months, as clinically indicated. Patients undergo PET at screening and treatment failure, and blood sample collection throughout the study. Patients may also undergo MRI as clinically indicated at screening and treatment failure.

After completion of study treatment, patients follow up at 3 months, 12 months, annually until year 5, and then optionally and per physician guidance every other year until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed prostate adenocarcinoma at the time of surgery
* Pathologic stages T2-T3b, Nx or N0-1, M0-1 as staged by the pathology report (American Joint Committee on Cancer [AJCC] Criteria 8th edition [Ed.])
* PSA post radical prostatectomy ≥ 0.1 and < 2.0 ng/mL ≤ 90 days prior to enrollment, obtained ≥ 6 weeks after surgery
* Eastern Cooperative Oncology Group (ECOG) performance status 0, 1, or 2 assessed ≤ 90 days of enrollment
* Patients must sign institutional review board (IRB) approved study specific informed consent
* Patients must complete all required pre-entry tests within the specified time frames
* Patients must be able to start treatment (ADT or radiation) ≤ 120 days of study registration
* Patients must be ≥ 18 years old
* Prostate cancer up to oligometastatic disease, up to 5 sites

Exclusion Criteria:

* Previous pelvic radiation
* Prior androgen deprivation therapy for prostate cancer and PSA ≥ 0.1 ng/mL
* Active rectal diverticulitis, Crohn's disease affecting the rectum, or ulcerative colitis (non-active diverticulitis and Crohn's disease not affecting the rectum are allowed)
* Prior systemic chemotherapy for prostate cancer
* History of proximal urethral stricture requiring dilatation
* Major medical, addictive, or psychiatric illness which in the investigator's opinion, will prevent the consent process, completion of the treatment and/or interfere with follow-up. (Consent by legal authorized representative is not permitted for this study)
* History of myocardial infarction or decompensated congestive heart failure (CHF) within the last 6 months
* On a transplant list
* More than oligometastatic disease > 5 metastatic sites

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2024-01-22 (Actual); Primary Completion 2030-01-22 (Estimated); Study Completion 2030-01-22 (Estimated)

PRIMARY OUTCOMES:
Incidence of grade 3 or higher genitourinary (GU)/gastrointestinal (GI) radiation treatment-related adverse events | Up to 2 years
  Defined as the proportion of patients experiencing an increase in GU/GI Common Terminology Criteria for Adverse Events version 5.0 to grade 3+ compared to pre-radiation therapy GU/GI toxicity over the number of patients eligible for toxicity evaluation at 2 years from the start of radiation therapy. This endpoint will be compared between patients treated with stereotactic body radiation therapy and hypofractionated radiation therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos E. Vargas, MD, Principal Investigator — Mayo Clinic
Locations (6):
- United States (6):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic Health System in Albert Lea, Albert Lea, Minnesota
  - Mayo Clinic Health System - Mankato, Mankato, Minnesota
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Mayo Clinic Health System-Eau Claire Clinic, Eau Claire, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials